CLINICAL TRIAL: NCT01293890
Title: Adherence to Medication and Its Impact on COPD Exacerbations: The AMICE Prospective Study
Brief Title: Adherence to Medication and Its Impact on Chronic Obstructive Pulmonary Disease (COPD) Exacerbations: The AMICE Prospective Study
Acronym: AMICE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: KU Leuven (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Marc Decramer, Prof. Dr., KU Leuven
Other Study IDs: B322201110500
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: adherence; medication; exacerbations; hospital admission
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- COPD patients with hospital admission for exacerbation

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) represents one of the most challenging chronic diseases of the 21st century: it is expected to be the fourth leading cause of death by 2030. COPD is characterized by pulmonary and extra-pulmonary systemic manifestations caused by partly irreversible expiratory airflow obstruction. The cornerstone of COPD management is the prescription of single or combined inhalation therapy, such as short- and long-acting bronchodilators, inhaled corticosteroids to possibly prevent disease progression, preserve lung function, relieve respiratory symptoms and prevent or treat exacerbations. Given the complex and lifelong treatment, one can expect that adherence to the prescribed inhalation therapy is not self-evident. Adherence can be defined as the "the extent to which a person's behaviour (taking medications, following a recommended diet and/or executing life-style changes) corresponds with the agreed recommendations of a health care provider". Inhaled medications have an additional complexity in that patients who intend to be adherent may be take the inhaled medication incorrectly, prohibiting proper therapeutic action. Taking less than the prescribed amount of medication, missing doses or stopping treatment for brief or extended periods will put the patient at risk for suboptimal disease control. Hence, the effectiveness will largely depend on the patient's ability to manage their disease adequately in daily life.

Using electronic monitoring, 3 studies in COPD found a prevalence of medication non-adherence of 51% which was worse than the average prevalence of 29% (range 3-66%) found across diseases such as hypertension, cancer, epilepsia, infections and HIV.

The existing evidence on risk factors for nonadherence in COPD is mostly anecdotic and not guided by behavioral models. According to the integrated model of behavioral prediction (IMBP), barriers, skills and ability and intention are the most important drivers of adherence (i.e. medication adherence).

The aims of the study are the following:

* To prospectively investigate the impact of medication nonadherence on time to exacerbation (primary end-point) and exacerbation rate, FEV1, hospitalization rate and duration, and quality of life (secondary end-points) at 1 year follow-up using electronic monitoring
* To investigate risk factors for medication nonadherence, using the Integrated Model of Behavioral Prediction as a theoretical framework
* To determine the diagnostic accuracy of different measures of medication nonadherence (i.e. pill count, self-report and physician rating) relative to electronic monitoring.
* To investigate the prevalence of nonadherence to other aspects of the therapeutic regimen, i.e. the use of concomitant medications, smoking cessation, alcohol use, physical activity, attendance to rehabilitation sessions and dietary adherence, their interrelations, and impact (alone and in combination) on time to first exacerbation.
* To investigate the interrelations in adherence to the various components of the therapeutic regimen.
* To investigate the impact of nonadherence to the other components of the therapeutic regimen (alone and in combination) on clinical outcomes (i.e. time to exacerbation, exacerbation rate/PPY, FEV1, hospitalization rate and duration, and quality of life at 1 year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of COPD
* Age > 40 years old
* Documented spirometry within the last 12 months with a post-bronchodilator FEV1 < 80% of predicted and an FEV1 < 70% of FVC (4 puffs of salbutamol 30 minutes prior to spirometry)
* Patients being hospitalized for an exacerbation at the University Hospitals of Leuven at time of enrollment
* Patients currently treated with Spiriva for at least 4 weeks at the start of the data collection (i.e. 4 weeks after hospitalization for an exacerbation)
* Oral fluency in Dutch
* Being capable to provide informed consent

Exclusion Criteria:

* A documented history of asthma or another respiratory disease
* An expected life expectancy of < 6 months
* Cognitive impairment (Mini Mental State Examination test results < 25) or presence of other co-morbidities preventing patients from completing the self-report instruments and/or using electronic monitoring
* Institutionalized patients, patients living in a nursing home or patients not managing their medications independently

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients that are admitted to the Pneumology of Geriatry Service of UZ Leuven after entering the emercency ward with a COPD exacerbation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-03; Primary Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
time to exacerbation | 1 year

SECONDARY OUTCOMES:
exacerbation rate | 1 year
Forced expiratory volume in one second (FEV1) | 1 year
Number of hospitalization rate due to exacerbations | 1 year
Duration of hospitalizations due to exacerbations | 1 year
Functional status | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Marc Decramer, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospital Leuven, Leuven, Flanders, Belgium